CLINICAL TRIAL: NCT02282501
Title: Leptin and Ghrelin in ICU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: özgür yağan (Other)
Responsible Party: Sponsor-Investigator, özgür yağan, MD, assistant professor, Ordu University
Organization: Ordu University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Odu-4
Record Dates: First submitted 2014-10-30; First posted 2014-11-04 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Critically Ill
Keywords: leptin levels; ghrelin levels
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- intermittent feeding (Active Comparator): Bolus infusion - The total daily feeding period was also 4-6 times a day.
  Interventions: Other: enteral feeding by nasogastric tube.
- continuous feeding (Active Comparator): Continuous infusion - The daily desired amount was offered continuously for 20 hours a day.
  Interventions: Other: enteral feeding by nasogastric tube.

INTERVENTIONS:
Other: enteral feeding by nasogastric tube. — method of administration enteral feeding by nasogastric tube.

SUMMARY:
Enteral alimentation is the preferred modality of support in critical patients who have acceptable digestive function and are unable to eat orally, but the advantages of continuous versus intermittent administration are surrounded by controversy.

This prospective, randomised study was designed to compare two enteral feeding methods with respect to changes in levels of leptin and ghrelin in ICU.

ELIGIBILITY:
Inclusion Criteria:

* who were unable to ingest an oral diet
* given decision on enteral feeding

Exclusion Criteria:

* Carcinomatosis
* irreversible coma
* death or discharge before 14 days of observation
* contraindication to enteral feeding
* intolerance to the prescribed nutrients or infusion regimen
* burn
* multiple trauma
* morbid obesity
* end stage liver or renal or lung disease
* severe sepsis or septic shock
* patients with percutaneous endoscopic gastrostomy
* immunosuppressive drug use
* severe hemodynamic instability
* massive blood transfusion

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-08; Primary Completion 2015-10 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in serum leptin concentration at three weeks in ICU | first, 7th, 14th and 21th day
Change from baseline in serum ghrelin concentration at three weeks in ICU | first, 7th, 14th and 21th day in ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesiology and Reanimation Dept. Ordu University Training and Research Hospital, Altinordu, Ordu, Turkey (Türkiye)